CLINICAL TRIAL: NCT00280839
Title: A Double-Blind, Placebo-Controlled, 11-Week Trial of Topiramate as an Aid to Smoking Cessation
Brief Title: Safety and Efficacy Study of Topiramate to Aid in Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAPSS-298
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- topiramate (Active Comparator)
  Interventions: Drug: Topiramate
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate
  Arms: topiramate
Drug: Placebo
  Arms: placebo

SUMMARY:
The purpose of this research study is to determine if topiramate is safe and effective in the treatment of smoking cessation

DETAILED DESCRIPTION:
Cigarette smoking is a pernicious national and global public health problem.1, 2 Nearly 50 million Americans smoke cigarettes despite widely publicized and acknowledged health warnings and restrictions on public smoking. Smoking has been branded as the most important preventable cause of all deaths in the United States (US), and 45% of smokers will die of tobacco related disorders.3, 4 Tobacco dependence is mediated, in part, by the reinforcing effects of nicotine.5 According to the US Public Health Service Clinical Practice Guideline, Treating Tobacco Use and Dependence, every patient attempting to stop smoking should be offered pharmacotherapy for smoking cessation.6 Pharmacological treatment strategies have included nicotine replacement therapy (NRT (nicotine formulations)), antagonist therapy (mecamylamine), therapies to make nicotine intake aversive (silver acetate), non-nicotine medications that mimic some of nicotine's neurophysiological effects (antidepressants), and medications to block craving and withdrawal symptoms (nicotine formulations, antidepressants, clonidine). A number of drug therapies for smoking cessation have demonstrated some efficacy in facilitating smoking cessation. These include NRT using a variety of nicotine formulations (e.g., pill, gum, patch, etc.);7-14 combined nicotine replacement and mecamylamine;15 the antidepressants, bupropion SR,16-19 nortriptyline,19-21 doxepin,22 and fluoxetine;23, 24 the alpha2 agonist, clonidine;25-27 and the anxiolytic, buspirone.28 Among these agents, first-line pharmacotherapies approved by the US Food and Drug Administration (FDA) that include bupropion SR and various NRT products have been found to approximately double long-term abstinence rates compared with placebo.29-31 However, roughly 7 to 8 out of 10 individuals who use these medications do not achieve long-term abstinence. I n addition to the limitations of currently available treatments for smoking cessation, several other clinical factors complicate the treatment of nicotine dependence. First, patients with a history of major depressive disorder appear to have a lower likelihood of achieving sustained smoking abstinence and an increased risk of depressive symptom emergence than patients without a history of major depressive disorder.32-44 Second, the emergence of prominent mood symptoms associated with nicotine withdrawal (e.g., anxiety, dysphoric or depressed mood, insomnia, irritability, and restlessness) reduce the likelihood of abstinence.35, 37, 44 Third, appetite increases and weight gain are also components of nicotine withdrawal and have negative health consequences.30, 45 Activation of the mesocorticolimbic dopamine (DA) system has been implicated in the reinforcing and dependence-producing effects of nicotine.46, 47 However, attempts to ameliorate the symptoms of nicotine dependence/withdrawal using DA receptors as therapeutic targets has met with only modest success.48, 49 Recent studies in rodents suggest that glutamatergic activation of N-methyl-D-aspartate (NMDA) receptors within the ventral tegmentum (VT) may be needed for nicotine to stimulate dopamine release in the nucleus accumbens.50-52 These findings are consistent with the reduction of nicotine-induced increases in locomotor activity observed with microinfusion of ionotropic glutamate receptor antagonists.53, 54 Thus, agents that indirectly modulate dopaminergic neurotransmission in the mesocorticolimbic reward circuit via their effects on presynaptic glutamatergic inputs to these dopamine neurons offer promise as novel adjuvants in the treatment of nicotine addiction.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria before entering the study:

1. Subjects who are daily smokers and smoke an average of ≥10 cigarettes/day within the 2 months prior to Visit 1 (Day -7).
2. Subjects must score ≥6 on the Motivation Scale.
3. Subjects must have a BMI ≥18 kg/m2.
4. Subjects must be between 18 and 65 years of age, inclusive.
5. Subjects can be male or female and must be in generally good health as confirmed by medical history, baseline psychiatric history, physical examination, laboratory tests and vital signs.
6. Female subjects must be:

   * postmenopausal for at least one year, or
   * practicing an effective method of birth control (e.g., surgically sterile, prescription oral contraceptives, contraceptive injections, intrauterine device, spermicide with barrier, contraceptive patch, contraceptive ring, male partner sterilization, abstinence and agree to continue abstinence or to use an acceptable method of contraception, as listed above, should sexual activity commence) before entry and throughout the study; have a negative urine pregnancy test at Visit 1 (Day -7).
7. Subjects must be able to take oral medication, adhere to the medication regimens and be willing to return for regular visits. CAPSS-298 Amendment 2 9 April 7, 2004
8. Subjects must be able and willing to read written instructions and complete all scales and inventories required by the protocol.
9. Subjects must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Subjects who have a current or recent (within 12 months of Visit 2, Day 1) MINI diagnosis of substance dependence or abuse (with the exception of nicotine or caffeine dependence).
2. Subjects with any current Axis I psychiatric disorder as defined by DSM-IV-TR™ and supported by the MINI, other than nicotine dependence, that in the investigator's judgment might require intervention with either pharmacological or non-pharmacological therapy over the course of the study.
3. Subjects with a history of personality disorder (e.g., schizotypal or borderline) considered by the investigator to likely interfere with assessment or compliance with treatment.
4. Subjects who have begun to receive formal psychotherapy (cognitive-behavioral therapy, behavioral therapy, or self-guided cognitive-behavioral therapy), hypnosis, acupuncture, or other non-pharmacological therapy for smoking cessation or any other psychiatric disorder within 3 months prior to Visit 1 (Day -7). Note: Subjects who have been engaged in formal psychotherapy for treatment other than nicotine dependence for >3 months and plan to maintain therapy throughout the study will be considered on a case-by-case basis.
5. Subjects who have received a prohibited medication described in the Concomitant Therapy section of the protocol and who have not met the washout criteria specified in Attachment 1.
6. Subjects who are considered to represent a significant risk of suicidal or violent behavior in the judgment of the investigator.
7. Subjects with a positive urine drug screening [cocaine, amphetamines, tetrahydrocannabinol (THC), benzodiazepines and opiates] at Visit 1 (Day -7). Note: Subjects with a positive urine drug screen for THC may be retested in 7 days and enrolled if they a) continue to meet inclusion/exclusion criteria and b) have a negative urine drug screen upon retest.
8. Female subjects who are pregnant or lactating.
9. Subjects with a history of nephrolithiasis.
10. Subjects known to have clinically significant medical conditions, including but not limited to:

    * symptomatic coronary artery or peripheral vascular disease;
    * malignancy or history of malignancy within the past 5 years (except basal cell carcinoma);
    * renal disease and/or impaired renal function as defined by subjects with an estimated creatinine clearance of ≤60 mL/min; CAPSS-298 Amendment 2 10 April 7, 2004
    * diseases of the gastrointestinal system including active liver disease;
    * subjects with AST and/or ALT >2 times the upper limit of the normal range and/or serum bilirubin >2 times the upper limit of normal at Visit 1 (Day -7); Note: if these values are abnormal they can be retested prior to Visit 2 (Day 1). If the repeat study is within the limits of the protocol, the subject may be randomized.
    * pulmonary disorders including subjects with active tuberculosis;
    * endocrinological disorders;
    * neurological disorders including subjects with seizure disorders and subjects with progressive and degenerative neurological disorders (e.g., multiple sclerosis);
    * any disease or condition that compromises the function of those body systems that could result in altered absorption, excess accumulation or impaired metabolism or excretion of topiramate; or
    * subjects with myocardial infarction, unstable angina, stroke or other major cardiovascular event within 6 months of the screening period.
11. Subjects with prior non-response to topiramate for the treatment of smoking cessation following an adequate trial.
12. Subjects who have previously been treated with topiramate for any reason and discontinued treatment due to an adverse event or due to a hypersensitivity reaction to topiramate.
13. Subjects who in the opinion of the investigator should not be enrolled in the study because of the precautions, warnings or contraindications outlined in the topiramate package insert.
14. Subjects who are employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.
15. Subjects who are members of the same household.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Keck, Jr., MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Anthenelli RM, Blom TJ, McElroy SL, Keck PE Jr. Preliminary evidence for gender-specific effects of topiramate as a potential aid to smoking cessation. Addiction. 2008 Apr;103(4):687-94. doi: 10.1111/j.1360-0443.2008.02148.x. PMID 18339115